CLINICAL TRIAL: NCT06098092
Title: Experimental Validation of the Long-term Accuracy of Blood Pressure Measurement Using a Smartwatch
Acronym: BPLONG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Czech Technical University in Prague (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: NVT_02_2023
Record Dates: First submitted 2023-10-09; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Hypertension; Blood Pressure
Keywords: Smartwatch; Blood pressure; Heart rate
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Interventional prospective single-arm study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Long-term Blood pressure and Heart rate monitoring with reference digital tonometer and smartwatch (Experimental): Measurement of a non-invasive Blood pressure and Heart rate using a reference medical grade digital tonometer Omron and a smartwatch Samsung Galaxy Watch during 20-40 days every morning and evening.
  Interventions: Other: Long-term non-invasive Blood pressure monitoring

INTERVENTIONS:
Other: Long-term non-invasive Blood pressure monitoring — All measurements during the experiment include only non-invasive Blood pressure and Heart rate measurements. Measurements will be taken using a smartwatch attached to the wrist and a digital tonometer with a cuff placed on the other arm. Paired readings will be compared.
  Other Names: Long-term non-invasive Heart rate monitoring

SUMMARY:
The aim of the study is to perform an experimental validation of the long-term accuracy of blood pressure measurement using the Samsung Galaxy Smartwatch

DETAILED DESCRIPTION:
Blood pressure is one of the basic vital signs monitored and is one of the most important indicators of a patient's health status. Cardiovascular disease is one of the leading causes of death worldwide. One of the major risk factors for cardiovascular disease is hypertension, which is globally attributed to one third of deaths in the world population. To improve the prevention of hypertension, self-monitoring of blood pressure is increasingly recommended. This project involves an experimental validation of the long-term accuracy of blood pressure measurement using the Samsung Galaxy Smartwatch compared to a medical grade digital tonometer with a cuff placed on the arm.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteer

Exclusion Criteria:

* post-traumatic conditions of the upper limbs
* tattoos, birthmarks, injuries or diseases of the skin on the wrists of hands
* cardiac arrhythmias
* circulatory or peripheral varcular disease
* aortic valve disease
* myocardiopathy
* other cardiovascular diseases
* pregnancy
* kidney disease
* diabetes
* neurotic disorder
* haemostatic disorders
* use of blood-thinning drugs

Min Age: 22 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-10-13 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-10-15 (Estimated)

PRIMARY OUTCOMES:
Blood pressure agreement between smartwatch and digital tonometer | 20-40 days
  The agreement of Blood pressure measurements between smartwatch and medical grade reference digital tonometer

SECONDARY OUTCOMES:
Heart rate agreement between smartwatch and digital tonometer | 20-40 days
  The agreement of Heart rate measurements between smartwatch and medical grade reference digital tonometer

CONTACTS AND LOCATIONS:
Overall Officials: Jakub Rafl, Principal Investigator — Czech Technical University
Locations (1):
- Czech Technical University in Prague, Kladno, Czechia

IPD SHARING:
Plan to Share IPD: Yes
The measured data will be shared publicly in the data repository on web page: https://ventilation.fbmi.cvut.cz/data/
Time Frame: Unlimited from the time of processing complete measured data
Access Criteria: Publicly available to everyone
URL: https://ventilation.fbmi.cvut.cz/data/

REFERENCES:
- [Derived] Walzel S, Sebestova H, Rafl-Huttova V, Rozanek M, Rafl J. Long-term accuracy and stability of blood pressure measurements from a smartwatch: Prospective validation study. Digit Health. 2026 Jan 22;12:20552076261415923. doi: 10.1177/20552076261415923. eCollection 2026 Jan-Dec. PMID 41602947